CLINICAL TRIAL: NCT06234618
Title: Study of Visual Deprivation on EEG Signal in Stroke Patients
Brief Title: The Effect of Covered Eye Walking on Electroencephalogram in Stroke Patients Compared With Open Eye Walking
Status: Suspended | Type: Observational
Why Stopped: The researchers would like to conduct a larger study and cover the contents of this study.
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhao Jing, Junior physiotherapist, Nanjing Medical University
Other Study IDs: ZD2022065
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Electroencephalography; walking; visual deprivation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patients: Stroke patients who can walk without assistance in their daily life.
  Interventions: Other: visual deprivation

INTERVENTIONS:
Other: visual deprivation — A group of patients walking with eyes open and walking with visual deprivation.

SUMMARY:
Post-stroke walking abnormalities present significant rehabilitation challenges. Visual deprivation training has been shown to be more effective than open-eye training. The investigators intend to examine the changes in electroencephalography patterns in stroke patients during visually deprived walking tasks.

The stroke participants will be fitted with a brain cap. The participants will walk with their eyes open for 60 seconds, and then their eyes will be blindfolded as they continue walking for another 60 seconds. Electroencephalography will monitor the signals in real-time during both walks.

DETAILED DESCRIPTION:
The electroencephalography data collection will be conducted in the Rehabilitation Department of Geriatric Hospital Affiliated with Nanjing Medical University. Upon commencing the experiment, participants will walk at a comfortable pace with their eyes open for a duration of 60 seconds. Following this initial test, a rest period of five minutes will be provided. For the visual deprivation walking trial, participants will be instructed to keep their eyes open throughout the trial. Investigators will apply an adequately sized blindfold to ensure complete visual deprivation, and the participants will proceed to walk for 60 seconds. During both trials, one investigator will remain one step behind the participant at all times to ensure safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Disease duration of more than 14 days
* Ability to walk at least 10 m without assistance,

Exclusion Criteria:

* Visual impairment
* Severe cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients in a hospital inpatient unit
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
phase locking value | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  used to evaluate the phase synchronization relationship between two signals.
phase lag Index | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  evaluate the degree of phase synchronization and the symmetry of neural oscillatory

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li Zhang, doctor, Study Director — Geriatric Hospital of Nanjing Medical University
Locations (1):
- Geriatric Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Three months after publication.
Access Criteria: Request from the researchers by email.

REFERENCES:
- [Background] Oliveira AS, Schlink BR, Hairston WD, Konig P, Ferris DP. Restricted vision increases sensorimotor cortex involvement in human walking. J Neurophysiol. 2017 Oct 1;118(4):1943-1951. doi: 10.1152/jn.00926.2016. Epub 2017 Jul 5. PMID 28679843
- See also: In this paper, the electroencephalography changes of normal people during visual deprivation walking were studied — http://pubmed.ncbi.nlm.nih.gov/28679843/